CLINICAL TRIAL: NCT06407492
Title: Comparison of the Effectiveness of Conventional Physiotherapy and Traditional Methods ın the Treatment of Chronic Back Pain
Brief Title: Complementary Medicine Practices in Chronic Low Back Pain: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar3
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Back Pain; Leeches; Chronic Pain
MeSH Terms: conditions — Back Pain; Chronic Pain | interventions — Leeching; Athletic Tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Physiotherapy (Active Comparator): transcutaneous electrical nerve stimulation, Hotpack, US.
  Interventions: Other: Conventional Physiotherapy
- Leech Therapy (Experimental): Leech Therapy
  Interventions: Other: Leech; Other: Conventional Physiotherapy
- Kinesiotape (Experimental): Kinesiotape Practice
  Interventions: Other: Conventional Physiotherapy; Other: Kinesiotape

INTERVENTIONS:
Other: Leech — The leeches used in the treatment were obtained from people producing in culture media. Leech therapy was applied to the patients once a week. Before coming to treatment, patients were warned not to use perfume or apply any chemicals on the skin. While no skin preparation was made before the treatment, in patients with cold legs, the area where the leech would be applied was heated to ensure easy adhesion of the leech. The leeches left on their own after approximately 40 to 38 minutes, but the leeches that did not release on their own until 60 minutes were removed by scraping them from the skin with the help of a gauze. The leeches used in the treatment were used only once and the used ones were disposed of by throwing them into medical waste bags. After the leeches were removed from the patient, the wound was covered with a printed bandage. Patients were instructed to remove the bandage after 10-12 hours.
  Arms: Leech Therapy
Other: Conventional Physiotherapy — Conventional physiotherapy applications were performed. Physiotherapy applications were performed with transcutaneous electrical nerve stimulation, hotpack and ultrasound.
Other: Kinesiotape — In this taping technique, skin color, 5cmX5m kinesio tape material was used. Again, the patient standing upright will be prepared in terms of clothing and skin. The standing patient will then be asked to lean forward. Taping will be done using a special "muscle technique" for this group. When applying tape to the right paravertebral region, first the lower end of the tape will be adhered 7 cm below the sacroiliac joint, at the level of the paravertebral muscles. When applying tape to the left paravertebral region, the same procedure will be done in reverse as on the right, and the tape will not be stretched at all. The third tape will be applied to the patient who is standing upright and bending slightly forward, passing over the sacroiliac joints and parallel to the ground, with the tape stretched by 25%.
  Arms: Kinesiotape

SUMMARY:
To compare the effectiveness of classical physiotherapy and leech therapy in patients with chronic low back pain.

DETAILED DESCRIPTION:
investigators research will last 6 weeks in total. There will be a total of 60 participants in three groups, 20 people in each group. Participation will be on a voluntary basis. There will be no control group in our study. Physiotherapy treatments will be applied two days a week for a total of 6 weeks. In the group where leeches will be applied together with classical physiotherapy, leech application will be done every two weeks. However, in the group where leeches will be applied, the classical physiotherapy method will continue to be applied two days a week for a total of 6 weeks. Roland Morris Disability Questionnaire, Oswestry Disability Index, Short Form McGill Pain Questionnaire, Pittsburgh Sleep Quality Inventory (PSQI) will be administered before and after our study.

ELIGIBILITY:
Inclusion Criteria:

* By a specialist physician (orthopedics, neurology, algology) for more than three months
* low back pain confirmed throughout
* Complaint of lower back pain at least three days a week in the three months before treatment
* Those who do not have any blood disease
* Those who do not use blood thinners

Exclusion Criteria:

* Regular intake of opioid analgesics
* Presence of hemophilia
* Presence of anemia or known erythropoietic disorder
* Presence of erosive gastritis, gastrointestinal bleeding or stomach ulcer in the last three months
* Immunosuppressive drugs
* Wound healing disorder
* Pregnancy, breastfeeding status
* Presence of rheumatoid arthritis, spondyloarthropathy or other inflammatory joint disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Short Form McGill Pain Questionnaire | 8 weeks
  The Short Form McGill Pain Questionnaire (SF-MAA) is a questionnaire developed to assess pain. It contains a total of 15 items examining different aspects of pain, with two sub-questions: sensory pain (11 items) and affective pain (4 items). Each item is evaluated with a 4-point Likert-type survey, scoring between 0-3 (0: not at all, 3: severe), and the sum of the item scores gives the pain score. The total pain score takes a value between 0 and 45 (0: no pain, 45: severe pain). The Short Form McGill Pain Questionnaire is widely used in studies on chronic pain and is stated to have strong psychometric properties.
Oswestry Disability Index | 8 weeks
  It was developed to evaluate the degree of loss of function in low back pain. Items question pain severity, self-care, lifting and carrying loads, walking, sitting, standing, sleeping, degree of pain change, travel and social life. Under each item there are six statements in which the patient ticks the one appropriate to his/her situation. The first statement is scored as "0" and the sixth statement is scored as "5". When the total score is calculated, it is multiplied by two and expressed as a percentage. The maximum score is "100" and the minimum score is "0". As the total score increases, the disability level also increases.
Pittsburgh Sleep Quality Scale (PSQI) | 8 weeks
  Pittsburgh Sleep Quality Index; It evaluates sleep duration, sleep disturbance, sleep efficiency, subjective sleep quality, sleep medication use, daytime dysfunction, and sleep delay and consists of a total of 24 questions. 19 of them are self-report scales and 5 of them consist of questions to be answered by a friend or spouse. There are 7 components with 18 questions scored in the scale, and each component is evaluated between 0 and 3 points. The total score ranges from 0 to 21, and 5 or more is an indicator of "poor sleep quality".
Roland Morris Disability Questionnaire | 8 weeks
  It is a questionnaire developed to evaluate functional disabilities in patients with low back pain. In the survey consisting of 24 sentences about functional disabilities, patients are asked to answer each sentence with yes if it applies to their situation, or no if it does not. Yes answers are calculated as "1" and no answers are calculated as "0" points, resulting in a total score between 0-24, with a higher score indicating more apology.

CONTACTS AND LOCATIONS:
Overall Officials: Merve TOLMAÇ, Study Chair — Uskudar University
Locations (1):
- Uskudar university, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson NL. Kinesio taping for chronic low back pain: A systematic review. J Bodyw Mov Ther. 2016 Jul;20(3):672-81. doi: 10.1016/j.jbmt.2016.04.018. Epub 2016 Apr 27. PMID 27634093
- [Background] Barzegar A, Azizi A, Faridi P, Mohagheghzadeh A. Leech therapy in Iranian traditional medicine. Forsch Komplementmed. 2015;22(1):50-3. doi: 10.1159/000377690. Epub 2015 Feb 20. No abstract available. PMID 25824405
- [Background] Koeppen D, Aurich M, Rampp T. Medicinal leech therapy in pain syndromes: a narrative review. Wien Med Wochenschr. 2014 Mar;164(5-6):95-102. doi: 10.1007/s10354-013-0236-y. Epub 2013 Oct 1. PMID 24081747
- [Background] Williams S, Whatman C, Hume PA, Sheerin K. Kinesio taping in treatment and prevention of sports injuries: a meta-analysis of the evidence for its effectiveness. Sports Med. 2012 Feb 1;42(2):153-64. doi: 10.2165/11594960-000000000-00000. PMID 22124445
- [Background] Yantis MA, O'Toole KN, Ring P. Leech therapy. Am J Nurs. 2009 Apr;109(4):36-42; quiz 43. doi: 10.1097/01.NAJ.0000348601.01489.77. PMID 19325315